CLINICAL TRIAL: NCT03375255
Title: A Phase 1 Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Dose of SRP-5051 in Patients With Duchenne Muscular Dystrophy Amenable to Exon 51 Skipping Treatment
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of a Single Dose of SRP-5051 (Vesleteplirsen) in Patients With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5051-101
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne Muscular Dystrophy; Exon Skipping; DMD; Exon 51; Ambulatory; Pediatric; Nonambulatory; Peptide-conjugated phosphorodiamidate morpholino oligomer (PPMO); Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRP-5051 (Experimental): Patients will be sequentially assigned to receive 1 of the 5 escalating dose levels of SRP-5051 on Day 1.
  Patients who complete the study and continue to meet safety eligibility criteria will have the opportunity to enroll in an open-label extension study to continue to receive SRP-5051.
  Interventions: Drug: SRP-5051

INTERVENTIONS:
Drug: SRP-5051 — Single dose of SRP-5051 administered as an intravenous (IV) infusion.
  Other Names: vesleteplirsen

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of 5 escalating doses of SRP-5051 (vesleteplirsen) administered as a single dose to patients with DMD amenable to exon 51 skipping treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has a genetic diagnosis of DMD and an out-of-frame deletion mutation of the DMD gene amenable to exon 51 skipping treatment
* Has been on a stable dose of oral corticosteroids for at least 12 weeks prior to study drug administration with continued dosing of oral corticosteroids while participating in the study*, or has not received corticosteroids for at least 12 weeks prior to study drug administration and will not initiate dosing of oral corticosteroids while participating in the study

Exclusion Criteria:

* Has a left ventricular ejection fraction (LVEF) less than (<) 40 percent (%) based on an echocardiogram (ECHO) performed within 3 months prior to Screening or at the Screening visit
* Has a QT interval corrected with Fridericia's method (QTcF) >= 450 millisecond (msec) on the Screening electrocardiogram (ECG)
* Initiation or change of dosing (except for modifications to accommodate changes in weight) within 12 weeks prior to Screening and while participating in the study for any of the following: angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blocking agents (ARBs), beta-blockers, or potassium
* Requires antiarrhythmic and/or diuretic therapy for heart failure
* Forced vital capacity (FVC) <40% of predicted value within 3 months of Screening or at the Screening visit
* Known kidney disease or had an acute kidney injury within 6 months prior to Screening
* Treatment with eteplirsen or drisapersen within 6 months prior to Screening, or any experimental gene therapy for the treatment of DMD at any time
* Use of any herbal medication/supplement containing aristolochic acid

Other inclusion/exclusion criteria apply.

*The dose of steroids must remain constant except for modifications to accommodate changes in weight.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | From signing of informed consent to 12 weeks after the last infusion of SRP-5051 (Up to 14 weeks)
  An AE is any untoward medical occurrence in a clinical trial participant, which does not necessarily have a causal relationship with the investigational drug. An AE can, therefore, be any unfavorable and unintended symptom, sign, disease, condition, or test abnormality that occurs during or after administration of the study drug, whether or not considered related to the study drug.

SECONDARY OUTCOMES:
Maximum Plasma concentration (Cmax) of SRP-5051 | Pre-dose, mid-infusion, end of infusion, post-dose (0.25, 0.5, 1, 2, 4, 8, 12 hours)
  Plasma samples to be collected via peripheral venipuncture from the contralateral arm used for drug infusion.
Area under the plasma concentration versus time curve (AUC) of SRP-5051 | Pre-dose, mid-infusion, end of infusion, post-dose (0.25, 0.5, 1, 2, 4, 8, 12 hours)
  Plasma samples to be collected via peripheral venipuncture from the contralateral arm used for drug infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (8):
- United States (7):
  - Neuromuscular Research Center, Sacramento, California
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No